CLINICAL TRIAL: NCT04433806
Title: The Feasibility of Primary Care Referrals to Community-based Lifestyle Programs for Management of Obesity
Brief Title: Primary Care Referrals to Community-based Lifestyle Programs for Management of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tamim I. Rajjo, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-010206
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Lifestyle, Healthy; Community Based Programs; Primary Care Referrals
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 25 subjects, all referred to community based program for weight loss at ExercisAbilities
  Interventions: Behavioral: Referral to weight loss program

INTERVENTIONS:
Behavioral: Referral to weight loss program — 16 weeks Diabetes Prevention Program based weight loss program at a local community partner

SUMMARY:
The purposes of this study is to evaluate the feasibility of providing a community based referral to Mayo Clinic Employee and Community Health patients for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are between 18-65 years of age
* Patients who have a BMI between 25-39.9 kg/m2
* Ability to provide informed consent
* Ability to complete the Diabetes Prevention Program including dietary and physical activity recommendations
* Motivated to lose weight (assessed to be in the preparation or action stage)

Exclusion Criteria:

* Have used weight loss medications or participated in a weight loss program within the past 30 days.
* Are currently enrolled in DPP or other ExercisAbilities weight loss programs
* Are currently taking supplements known to affect weight.
* Have had weight fluctuations of 20 pounds or more in the past 6 months (EMR check and self-report)
* Have an active untreated clinically significant psychiatric condition (psychosis, bipolar disorder, or depression)
* Are currently pregnant or breastfeeding, or are of child-bearing potential and are likely to become pregnant during the study (within the next 4 months following enrollment)
* Have a history in the past 4 months of any major cardiovascular events including heart valve disease, cardiac arrhythmias, congestive heart failure, acute coronary syndrome, stroke, transient ischemic attack, or peripheral vascular disease
* Have current uncontrolled hypertension (systolic > 160 mm Hg or diastolic > 95 mm Hg) documented on 2 separate occasions
* Have clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, lymphatic, respiratory, or metabolic disease (such as diabetes) or active cancer or are within 1 year of cancer remission
* Have a known history of any condition or factor judged by the investigator/study team to preclude participation in the study or which might hinder adherence
* Have any co-morbidity that is deemed exclusionary at the discretion of the provider.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Participants recruited | Through study completion, approximately 28 weeks
  Total number of participants recruited
Participants enrolled | Through study completion, approximately 28 weeks
  Total number of participants enrolled
Participants accrued | Through study completion, approximately 28 weeks
  Total number of participants accrued
Participants to withdrawn or terminate study participation | Through study completion, approximately 28 weeks
  Total number of participants to withdrawn or terminate study participation

SECONDARY OUTCOMES:
Participant satisfaction | At study completion, approximately 28 weeks
  Measured using the self-reported Was It Worth It (WIWI) Questionnaire that uses a total of 13 questions that asks feedback on participants experience and satisfaction with the Mayo Clinic/ExercisAbilities weight loss program.
Staff satisfaction | At study completion, approximately 28 weeks
  Measured using the self-reported ExercisAbilities Staff Survey (Post-Intervention) that uses a total of 3 questions to rate experience on a scale of very satisfied to extremely not satisfied.
Change in weight | Baseline, week 16, week 28
  Change in participant's weight measure in kilograms (kg)
Change in Body Mass Index (BMI) | Baseline, week 16, week 28
  Change in participant's BMI calculated by weight in kilograms divided by the square of height in meters (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Rajjo, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials